CLINICAL TRIAL: NCT02917122
Title: The Therapeutic Effect of Transcranial Direct Current Stimulation on Depression in Parkinson's Disease
Acronym: Parkinson's
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding is insufficient.
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Kao Chin, Chen, assistant professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-103-079
Record Dates: First submitted 2016-06-30; First posted 2016-09-28 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease; Depression
Keywords: Parkinson disease; transcranial direct current stimulation; depression; dopamine transporter; single photon emission computerized tomography
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sertraline + sham tDCS (Placebo Comparator): Patients will take sham tDCS.
  Interventions: Drug: Sertraline; Device: sham tDCS
- sertraline + active tDCS (Active Comparator): Patients will take 12 tDCS sessions (30min for each session): first 10 consecutive sessions for two weeks (Monday to Friday), and then 2 follow-up sessions scheduled 2 and 4 weeks after the consecutive treatment.
  Interventions: Device: active tDCS; Drug: Sertraline

INTERVENTIONS:
Device: active tDCS — Patients will take 12 tDCS sessions (30min for each session): first 10 consecutive sessions for two weeks (Monday to Friday), and then 2 follow-up sessions scheduled 2 and 4 weeks after the consecutive treatment.
  Arms: sertraline + active tDCS
Drug: Sertraline — Patients will take Sertraline.
Device: sham tDCS — Patients will take 12 tDCS sessions (30min for each session): first 10 consecutive sessions for two weeks (Monday to Friday), and then 2 follow-up sessions scheduled 2 and 4 weeks after the consecutive treatment.
  Arms: sertraline + sham tDCS

SUMMARY:
Parkinson's disease (PD) is one of the most common neurological diseases manifested by movement disturbance. The concomitant psychiatric symptoms, especially depression, are often observed and have also great impact on patients' quality of life. The treatment of depressive symptoms in PD with antidepressants as the majority remains variable and inefficient, which complicates the disease prognosis. Transcranial direct current stimulation (tDCS) is a non-invasive brain modulation technique and has been demonstrated to improve psychiatric diseases such as major depression. In this study the investigators will assess the combined effects of tDCS on sertraline for the treatment of depression in PD. Ten sessions of tDCS in two weeks will be applied and the follow-up evaluation will continue bi-weekly for one month after completing all sessions. The efficacy of tDCS vs sertraline will be compared and evaluated with behavioral and cognitive outcome. In addition, the investigators will evaluate if the baseline dopaminergic activity in brain could predict the treatment outcome by using SPECT imaging. The investigators aim to establish the therapeutic parameters and safety criteria of tDCS as an add-on or alternative therapy, and further enhance the overall clinical efficacy in the treatment of depression in PD.

DETAILED DESCRIPTION:
Study design

This study is a factorial randomized, placebo-control trial, including 2 groups: 'sertraline only' (sertraline + sham tDCS), and 'combined treatment' (sertraline + active tDCS). It is planned to recruit 20 subjects for each group, which results in all together 40 participants. Patients will take 12 tDCS sessions (30min for each session): first 10 consecutive sessions for two weeks (Monday to Friday), and then 2 follow-up sessions scheduled 2 and 4 weeks after the consecutive treatment. Both pharmacological and tDCS intervention will be started simultaneously on the first day of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Suffers from Parkinson's disease fulfill the Parkinson's Disease Society Brain Bank clinical criteria with insidious 2 or more PD symptoms (bradykinesia, tremor, or rigidity).
4. Suffers from "DSM-IV major depressive disorder, single episode" or "DSM-IV major depressive disorder, recurrent" according to Diagnostic & Statistical Manual of Mental Disorders, 4th Edition - Text Revision (DSM-IV-TR) criteria.
5. Reported duration of the current episode is ≥4 weeks and has not been treated with antidepressants.
6. Has a Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≥20 at the screening (baseline) visit.
7. Is a man or woman aged 18 to 75 years, inclusive.

Exclusion criteria:

1. Subjects known to have allergies to sertraline and pimozide.
2. Subjects showed any signs of substantial risk of suicide during the trial.
3. Subjects ever received electroconvulsive treatment.
4. Subjects co-morbid with other major mental disorders or with substance/alcohol dependence or abuse in the past 6 months per DSM-IV criteria.
5. Nursing women, pregnant women or patients suspected pregnant.
6. History or presence of clinically significant hepatic, cardiovascular or renal disease, or other serious medical disease that might compromise the study.
7. History of seizure disorder or need to taking medications that increase the risk of seizure.
8. History or presence of dementia and any previous history of brain tumor, brain arteriovenous malformation, encephalitis or meningitis.
9. Subjects ever received or plan to receive brain surgery during the trial.
10. Subjects with pacemaker or are contraindicated for MRI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kao Chin Chen, PhD, Study Chair — National Cheng-Kung University Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sertraline + Sham tDCS | Sertraline + Active tDCS
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline + Sham tDCS | Sertraline + Active tDCS | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.00 (8.50) | 61.86 (9.82) | 61.93 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change of Modified-Unified Parkinson's Disease Rating Scale Among Different Weeks
Description: mds: modified-Unified Parkinson's Disease
  mds1 non-motor experiences of daily living: summed, 0-52 mds2 motor experiences of daily living: summed, 0-52 mds3 motor examination: summed, 0-132 mds4 motor complications: summed, 0-24
  higher value is worse
Time Frame: week 0 and 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline + Sham tDCS | Sertraline + Active tDCS
Number analyzed (Participants) | 6 | 4
score on a scale
  mds1 non-motor experiences of daily living-week0 | 9.00 (5.48) | 10.00 (4.83)
  mds1 non-motor experiences of daily living-week6 | 6.17 (3.43) | 8.25 (3.10)
  mds2 motor experiences of daily living-week0 | 5.33 (3.50) | 2.25 (2.06)
  mds2 motor experiences of daily living-week6 | 2.17 (1.33) | 4.75 (3.20)
  mds3 motor examination-week0 | 23.50 (12.93) | 18.75 (6.40)
  mds3 motor examination-week6 | 22.17 (10.34) | 19.50 (5.00)
  mds4 motor complications-week0 | 0.50 (1.22) | 2.75 (3.77)
  mds4 motor complications-week6 | 1.00 (1.55) | 1.25 (2.50)

2. Primary Outcome: Change of Hamilton Rating Scale for Depression Among Different Weeks
Description: Hamilton Rating Scale for Depression: summed, 0-50
  higher value is worse
Time Frame: week 0 and 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline + Sham tDCS | Sertraline + Active tDCS
Number analyzed (Participants) | 5 | 6
score on a scale
  week0 | 21.83 (4.79) | 27.40 (4.22)
  week6 | 5.83 (4.36) | 10.20 (7.69)

3. Primary Outcome: Change of Taiwanese Depression Questionnaire Among Different Weeks
Description: Taiwanese Depression Questionnaire: summed, 0-54
  higher value is worse
Time Frame: week 0 and 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sertraline + Sham tDCS | Sertraline + Active tDCS
Number analyzed (Participants) | 6 | 5
score on a scale
  week0 | 25.50 (11.64) | 24.80 (11.19)
  week6 | 14.83 (12.34) | 18.60 (16.01)

ADVERSE EVENTS:
Time Frame: week -1, 0, 2, 4, 6
Arm/Group | Sertraline + Sham tDCS | Sertraline + Active tDCS
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT02917122/Prot_SAP_ICF_000.pdf